CLINICAL TRIAL: NCT03282201
Title: The Effect of Blood Transfusion on Recovery After Major Arthroplasties
Brief Title: A Survey on Blood Transfusions in Major Artrhoplasty Operations
Status: Completed | Type: Observational
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Associate Proffesor, Diskapi Teaching and Research Hospital
Other Study IDs: TransfusionArthroplasty
Record Dates: First submitted 2017-09-12; First posted 2017-09-13 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2017-09

CONDITIONS: Arthropathy of Hip; Arthropathy of Knee
MeSH Terms: interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfused: Patients in whom blood transfusion is used
  Interventions: Other: Transfusion
- Nontransfused: Patients in whom blood transfusion is not used

INTERVENTIONS:
Other: Transfusion — Transfusion of red blood cells, fresh frozen plasma, platelets
  Groups: Transfused

SUMMARY:
The rate of hip, knee arthroplasties and their revision are increasing every year. The incidence of blood transfusion in these operations are reported 18%, 68%, and 39%, 67%, respectively. Blood transfusion is known to increase the risk of pulmonary, septic, wound and thromboembolic complications and is related to mortality. Restrictive transfusion protocols has cost-effective results in terms of reducing these complications, promoting early discharge and reduced frequency of re-admission.

Within this context, we aimed to evaluate the transfusion practice in our hospital, define the transfusion indicators and compare the transfused and non transfused patients in terms of recovery.

DETAILED DESCRIPTION:
After obtaining ethical approval Patients undergoing hip or knee arthroplasty or revision arthroplasty will be included in this prospective observational study.

Patient characteristics (age , gender, body mass index, ASA physical status, anticoagulant medication) Preoperative: hemoglobin, hematocrit, platelet, INR, APTT, PT values, the precence of preoperative anemia, anemia treatment modalities will be recorded.

Intraopreative: type and duration of surgery, anesthesia method, monitoring methods used, the amount of intraoprative adminestred fluids (crystalloid-colloid), amount of hemorrhage Postoperative: hemoglobin-hematocrit-platelet leve The amount of blood transfusion and the product used (erythrocyte suspension, fresh frozen plasma, thrombocyte-fibrinogen-factor concentration-cryoprecipitate-other ) Hemoglobin-hematocrit-platelet level before and after transfusion Indications for transfusion; hemoglobin threshold / physiological transfusion indicator; tachycardia, hypotension, low flow rate, desaturation, low SvO2, inotropic requirement, etc. / comorbidities / monitorisation findings, other, Discharge time of patients Early upright position (postoperative 2nd day), information on walking capacities (TUG - The Time Up and Go test) will be recorded and compared between transfused and non-transfused patients

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing major atrhroplasty

Exclusion Criteria:

* Pediatric patients

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major atrhroplasty
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-06-20 (Actual)

PRIMARY OUTCOMES:
Discharge time | Postoperative day 1-6 days
  Discharge time from hospital
TUG test | Postoperative day 1-2
  Walking without help

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Yazicioglu, Assoc Prof, Principal Investigator — Ministry of Health
Locations (1):
- Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Poitras S, Wood KS, Savard J, Dervin GF, Beaule PE. Predicting early clinical function after hip or knee arthroplasty. Bone Joint Res. 2015 Sep;4(9):145-51. doi: 10.1302/2046-3758.49.2000417. PMID 26336897
- [Background] Cram P, Vaughan-Sarrazin MS, Wolf B, Katz JN, Rosenthal GE. A comparison of total hip and knee replacement in specialty and general hospitals. J Bone Joint Surg Am. 2007 Aug;89(8):1675-84. doi: 10.2106/JBJS.F.00873. PMID 17671004
- [Result] Engoren M, Mitchell E, Perring P, Sferra J. The effect of erythrocyte blood transfusions on survival after surgery for hip fracture. J Trauma. 2008 Dec;65(6):1411-5. doi: 10.1097/TA.0b013e318157d9f9. PMID 19077635
- [Result] Kotze A, Carter LA, Scally AJ. Effect of a patient blood management programme on preoperative anaemia, transfusion rate, and outcome after primary hip or knee arthroplasty: a quality improvement cycle. Br J Anaesth. 2012 Jun;108(6):943-52. doi: 10.1093/bja/aes135. PMID 22593128